CLINICAL TRIAL: NCT06876974
Title: Assessment of Prognosis and Myocardial Reperfusion in Patients with ST-segment-elevation Myocardial Infarction (STEMI) According to Coronary Atherosclerotic Burden.
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Batric POPOVIC, Professor, Central Hospital, Nancy, France
Other Study IDs: 2025PI034
Record Dates: First submitted 2025-02-21; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: STEMI - ST Elevation Myocardial Infarction (MI)
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In the current literature, it has been widely demonstrated that the extend of coronary atherosclerotic burden is associated with adverse long-term outcomes. Little is known about the impact of atheroma burden and either myocardial reperfusion and short-term outcomes after ST-segment elevation myocardial infarction (STEMI). Several angiographic scores have been used to measure the extend and severity of coronary atheroma. The SYNTAX score and the Gensini score have been shown to be independent predictors of cardiovascular events and mortality in stable coronary artery disease as well as in myocardial infarction.

This research therefore aims to assess the impact of overall coronary atherosclerotic burden, measured by two angiographic scores (SYNTAX score and Gensini score), both before and after primary percutaneous angioplasty, in patients with STEMI according to different clinical subgroups.

ELIGIBILITY:
Inclusion criteria:

- patients presenting with STEMI and treated with primary PCI (pPCI) at the University Hospital of Nancy between 2003 and 2023.

Exclusion criteria:

- patients with missing or incomplete coronary angiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with STEMI and treated with primary PCI (pPCI) at the University Hospital of Nancy between 2003 and 2023.
  STEMI was defined as follows:
  1. continuous chest pain lasting at least 20 min
  2. ST-segment elevation ≥1 mm in ≥2 contiguous leads on a 12-lead electrocardiogram or left bundle branch block and (3) treatment within 24 h of pain onset.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 2 years
  all-cause mortality at 45 days, 1 year and 2 years
Recurrent acute coronary syndrome | 1 year
  Recurrent acute coronary syndrome at 1-year

SECONDARY OUTCOMES:
All-cause mortality in patients with STEMI related to out-of-hospital cardiac arrest or cardiogenic shock | 2 years
  All-cause mortality at 45 days, 1 year and 2 years in patients with STEMI related to out-of-hospital cardiac arrest or cardiogenic shock
Recurrent acute coronary syndrome in patients with STEMI related to out-of-hospital cardiac arrest or cardiogenic shock | 1 year
  Recurrent acute coronary syndrome at 1 year in patients with STEMI related to out-of-hospital cardiac arrest or cardiogenic shock

IPD SHARING:
Plan to Share IPD: Undecided